CLINICAL TRIAL: NCT00832195
Title: Footwear Prevention Study: Investigating the Effects of Running Shoe Pronation Control on the Risk of Injury
Brief Title: Footwear and Injury Prevention Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H08-02995
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Pronation Control
Keywords: running; injury; pronation; footwear.
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Footwear with motion controlling elements built into construction in order to reduce pronation of the foot and ankle during running.
  Interventions: Device: Motion Controlling Running Shoe
- 2 (Active Comparator): Footwear with standard neutral stabilization elements for the foot and ankle during running.
  Interventions: Device: Neutral Running Shoe

INTERVENTIONS:
Device: Motion Controlling Running Shoe — Running shoe with thermoplastic mid-foot shank stiffener, denser durometer foam on medial aspect of mid-sole, reinforced heel counter, wider sole-plate, and lateral foam crash-pad.
  Arms: 1
Device: Neutral Running Shoe — Standard running shoe with single density mid-sole foam.
  Arms: 2

SUMMARY:
The purpose of this study is to assess whether shoes that are more controlling for movement of the foot and ankle, compared to shoes that are less controlling, will reduce the overall number and severity of injuries experienced during a 13-week running programme. Our hypothesis is that runners who wear more controlling footwear during the 13-week programme will experience less injury events.

DETAILED DESCRIPTION:
The proposed study will be a non-blinded prospective randomized cohort design.

Subjects will include adult runners of both genders with no history of injury in the 6 months prior to study enrollment. Eligible participants will have no history of surgery or trauma to the lower extremity that might compromise their walking or running gait, and all subjects must be able to comfortably fit into their selected footwear.

Three different foot posture sub-group classifications will be recruited: neutral, mild to moderate, and excessive. The subjects' foot posture will be classified using the Foot Posture Index (Redmond et al. (2006)(1). Twenty four subjects are estimated to be required within each foot posture sub-group; therefore 72 subjects will be our goal for enrollment. Subjects within each foot posture sub-group will be randomized into one of two separate footwear conditions: both the neutral group and the mild to moderate pronator group will be divided to receive either a neutral cushioned running shoe (a.k.a. 'neutral shoe'), or a shoe with mild stability components for controlling overpronation (a.k.a. 'stability shoe'); participants in the excessive pronator sub-group will be randomized to receive either a 'stability shoe' or a shoe will aggressive motion controlling features (a.k.a. 'motion control shoe').

All subjects will undergo an initial baseline test, including an entrance interview for participant eligibility, training history, running injury history and documentation of lower extremity anthropometry (i.e. arch height, knee alignment, standing rearfoot position). Subjects will be randomized during their baseline test to their shoe condition and receive their shoes, training diary and running programme at that time.

Once all subjects have completed their baseline testing, the official running clinic start date will commence on the following Saturday. A running clinic is established so that all subjects will have a chance to meet together, along with knowledgeable run leaders and a study co-investigator (MR), in order to increase group cohesion and provide an opportunity for data monitoring, programme feedback and subject questions. All subjects will begin the running programme at the official running clinic start date. The programme is designed to prepare individuals for a half-marathon (21 kilometre) running event in 13 weeks. Subjects will run on their own time, as indicating in their running programme, for the rest of the week until meeting again the following Saturday. This schedule will be repeated for the entire 13 week duration of the programme.

Outcome variables of interest in this study include: 1) number of injury events, defined as a missed run workout that is associated with running related pain; 2) McGill Pain Questionnaire score(2) ; and 3) Visual Analog Scale (VAS) items for pain at rest, activities of daily living, during or immediately after running, respectively(3) . Outcome variables will be assessed at baseline, at the 6 week point in the running programme, and at the conclusion to the running programme.

All data will be entered into a spreadsheet and statistical analysis software package JMP Version 4.0.0 (SAS Institute Inc., Cary, NC). In calculating statistical power for subject recruitment, a 20% difference in the VAS pain scores across groups will be considered to be a clinically meaningful difference. Accordingly, assuming a standard deviation of 2.3 in the VAS scores, an alpha of 5% and a beta error-level of 10%, twenty four subjects will be required within each foot posture sub-group; therefore 69 subjects will be our goal for enrollment. Each foot posture sub-group will undergo its own analysis procedure. Levene's test of equality of variance will precede a factorial analysis of variance in determining whether there are significant main effects for time and footwear condition, as well as an interaction effect, for all three dependent (or outcome) variables. Alpha will be set at 0.05 for this study.

1. Redmond AC, Crosbie J, Ouvrier RA. Development and validation of a novel rating system for scoring standing foot posture: The Foot Posture Index. Clin Biomech 2006;21:89-98.
2. Melzack R. The McGill Pain Questionnaire: Major properties and scoring methods. Pain. 1975; 1: 277-299.
3. Wewers M.E. & Lowe N.K. A critical review of visual analogue scales in the measurement of clinical phenomena. Research in Nursing and Health 1990;13: 227-236.

ELIGIBILITY:
Inclusion Criteria:

* Adult, runner.

Exclusion Criteria:

* Not currently injured,
* No history of surgery to the lower extremity.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Injury status, as measured at baseline, 6 weeks, and at the end of the 13-week programme | 13 weeks

SECONDARY OUTCOMES:
Pain levels, as measured at baseline, 6 weeks, and at the end of the 13-week programme | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jack Taunton, MD, Principal Investigator — University of British Columbia; Michael Ryan, Study Director — University of British Columbia
Locations (1):
- Lady Sport, Vancouver, British Columbia, Canada